CLINICAL TRIAL: NCT06908655
Title: Diffusion Endometriosis MRI to Detect and Quantify Symptomatic Neurological Impairment in Pelvic Endometriosis
Acronym: TENDANSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Imagine Institute (Other); Sauver la vie Fundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP241481; 2024-A00538-39 (Other: Agence nationale de sécurité du médicament et des produits de santé); 24.05788.000362 (Other: Commission Nationale des Recherche Impliquant la Personne Humaine)
Record Dates: First submitted 2025-03-13; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-02

CONDITIONS: Endometriosis
Keywords: endometriosis; tractography; pelvic nervous tract
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-randomized, multicenter, diagnostic study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with symptoms compatible with possible endometriosis (Experimental): Patients will have an initial gynecological surgery consultation to determine the indication for MRI to diagnose and/or assess pelvic endometriosis. MRI will be performed at the HEGP, comprising a T2-weighted isotropic thin-section (3D) cube sequence (1 mm3), and a T1-weighted isotropic 3D DIXON sequence (1 mm3), for a total duration of 20 minutes (including set-up). Patients will also have a pelvic ultrasound if they have not already had one at a center specializing in endometriosis.
  They will have a further consultation after the MRI, so that the gynecological surgeon can discuss therapeutic management. All these procedures are performed as part of routine management.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — The procedure to be investigated will be to perform a diffusion tensor sequence during the MRI indicated as part of the treatment. The diffusion tensor sequence takes 10 minutes to acquire, for a total examination time of 30 minutes instead of 20 minutes, including set-up.

SUMMARY:
This research focuses on evaluating the ability of diffusion tensor imaging (DTI) to detect nerve damage in pelvic endometriosis. The primary objective is to visualize pelvic nerve plexuses to better understand the mechanisms of endometriosis-related neuropathic pain. Secondary objectives include comparing nerve damage between women with and without endometriosis.

To answer this question, it is planned to include 110 women with symptoms compatible with endometriosis, in Paris hospitals (Hôpital Cochin and HEGP). This research is funded by Assistance Publique - Hôpitaux de Paris. The expected duration of the research is 2 years, with individual participation of 3 months.

The research process will be as follows:

* Visit 0 (V0): Initial consultation to assess your state of health, complete pain questionnaires (EHP5, EHP30, DN4, EVA), and obtain your informed consent. Prescription of MRI.
* Visit 1 (V1): MRI with diffusion tensor imaging (DTI) within 60 days of V0. The MRI examination will be 10 minutes longer than the usual MRI. An intramuscular injection of glucagon hydrochloride will be given as part of the treatment.
* Visit 2 (V2): Follow-up consultation at 3 months, where the results of the standard MRI sequences will be discussed.

Research constraints and modalities:

* The addition of the DTI sequence extends the routine MRI by 10 minutes.
* You must attend each scheduled appointment. If you are unable to attend, please inform your doctor.
* No additional medications, treatments or samples are required for this study. You will be expected to follow your usual endometriosis treatments, with no specific restrictions on the drugs used, but please report any use of alternative medicine to your doctor.

No additional hospitalization is planned.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years
* Non-menopausal (menopause defined as absence of menstrual periods for 12 consecutive months)
* Referred to the department for clinical suspicion of endometriosis on questioning Or known endometriosis
* Requiring specialized MRI by a specialist in endometriosis and adenomyosis imaging for diagnosis or follow-up of endometriosis.
* Patient affiliated to social security
* Patient with signed informed consent
* Patient with a good understanding of the French language

Exclusion Criteria:

* Pregnant or breast-feeding women
* Contraindication to MRI: ocular metallic foreign body, pacemaker, mechanical heart valve, old vascular clips on cerebral aneurysm;
* Claustrophobic patients
* Contraindication to glucagen injection (anti-peristaltic);
* Previous pelvic surgery;
* Patient having participated in a therapeutic clinical trial involving a new molecule within 30 days prior to inclusion;
* suffering from a severe chronic disease (cancer, HIV, renal failure, ongoing liver or biliary disorders, chronic inflammatory digestive disease, arthritis or other chronic respiratory disorders) or gastrointestinal disorders deemed incompatible with the conduct of the study by the investigator;
* Vulnerable patients (legal protection, guardianship, curatorship);
* Patients receiving State Medical Aid.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
At least one measurable parameter (yes/no) on tractography in patients with or without endometriosis. | 3 months
  Evaluate the ability of the diffusion tensor sequence to visualize normal or pathological pelvic nerve plexuses (hypogastric and sciatic) in pelvic endometriosis. These parameters will be measured on MRI tractography images.
Proportion of patients with at least one relevant parameter evaluated by MRI-based tractography, in patients with or without endometriosis | Between 7 and 60 days after inclusion
  Number of patients (with or without endometriosis) in whom at least one parameter could be evaluated, divided by the total number of patients (with or without endometriosis) who attended an MRI-based tractography.
  Parameters expected to be evaluable with MRI-based tractography:
  * total volume
  * lengths
  * number of branches
  * tortuosity MRI will be exploited by independant readers, blinded from patients'clinical characteristics and diagnosis

SECONDARY OUTCOMES:
Proportion of patients with an individual relevant parameter evaluated by MRI-based tractography, in patients with or without endometriosis | Between 7 and 60 days after inclusion
  Number of patients (with or without endometriosis) in whom the individual parameter could be evaluated, divided by the total number of patients (with or without endometriosis) who attended an MRI-based tractography.
  Individual parameters expected to be evaluable with MRI-based tractography:
  * total volume
  * lengths
  * number of branches
  * tortuosity
Total volume evaluated by MRI-based tractography | Between 7 and 60 days after inclusion
  MRI stands for "Magnetic Resonance Imaging".
  In patients with vs without endometriosis: comparisons between patients with vs without endometriosis.
  In patients with endometriosis: comparisons according to (i) presence of endometriosis lesions (yes vs no), (ii) pain type (neuropathic vs other), (iii) endometriosis phenotype (endometriom vs deep endometriosis), (iv) localisation of lesions (pelvic wall vs sacro-rectus-genitourinary blade vs iliac incisure), all subgroups evaluated at inclusion.
Length of branches evaluated by MRI-based tractography. | Between 7 and 60 days after inclusion
  MRI stands for "Magnetic Resonance Imaging".
  In patients with vs without endometriosis: comparisons between patients with vs without endometriosis.
  In patients with endometriosis: comparisons according to (i) presence of endometriosis lesions (yes vs no), (ii) pain type (neuropathic vs other), (iii) endometriosis phenotype (endometriom vs deep endometriosis), (iv) localisation of lesions (pelvic wall vs sacro-rectus-genitourinary blade vs iliac incisure), all subgroups evaluated at inclusion.
Number of branches evaluated by MRI-based tractography. | Between 7 and 60 days after inclusion
  MRI stands for "Magnetic Resonance Imaging".
  In patients with vs without endometriosis: comparisons between patients with vs without endometriosis.
  In patients with endometriosis: comparisons according to (i) presence of endometriosis lesions (yes vs no), (ii) pain type (neuropathic vs other), (iii) endometriosis phenotype (endometriom vs deep endometriosis), (iv) localisation of lesions (pelvic wall vs sacro-rectus-genitourinary blade vs iliac incisure), all subgroups evaluated at inclusion.
Tortuosity evaluated by MRI-based tractography. | Between 7 and 60 days after inclusion
  MRI stands for "Magnetic Resonance Imaging".
  In patients with vs without endometriosis: comparisons between patients with vs without endometriosis.
  In patients with endometriosis: comparisons according to (i) presence of endometriosis lesions (yes vs no), (ii) pain type (neuropathic vs other), (iii) endometriosis phenotype (endometriom vs deep endometriosis), (iv) localisation of lesions (pelvic wall vs sacro-rectus-genitourinary blade vs iliac incisure), all subgroups evaluated at inclusion.
Proportion of patients with nerve lesions, in patients with endometriosis | Baseline
  Qualitative assessment of the presence of
  * localised lesions
  * diffuse lesions along the plexus
Inter-reader reproductibilty of nerve lesions, in patients with endometriosis | Baseline
  Cohen's Kappa for reproducibility between 2 readers who performed the qualitative assessment of the presence of
  * localised lesions
  * diffuse lesions along the plexus
Fractional Anisotropy, in patients with vs without endometriosis | Between 7 and 60 days after inclusion
  Comparisons between patients with vs without endometriosis.
  Individual parameters :
  * mean diffusity
  * axial diffusity
  * radial diffusity
Scores at EHP5 Quality of Life questionnaires, in patients with endometriosis | Baseline
  EHP-5 stands for "Endometriosis Health Profiles in 5 items". The higher the worse between 0 and 100.
  Sum of answer at each item divided by the number of answered items. Individual item of the EHP-5.
Scores at EHP30 Quality of Life questionnaires, in patients with endometriosis | Baseline
  EHP-30 stands for "Endometriosis Health Profiles in 30 core-items". The higher the worse between 0 and 100.
  Sum of score at each scale divided by the number of answered scales. Individual score at each scale of the EHP-30.
DN4-based and visual analog scale for pain assessment, in patients with endometriosis | Baseline
  DN4 stands for " Douleur Neuropathique en 4 questions " or " Neuropathic pain in 4 questions ". The higher the worse between 0 and 10.
  VAS stands for "Visual Analog Scale". The higher the worse between 0 and 10. Score at each part of DN4 pain questionnaire.
  Score at part 4 on deep pain augmented by 3 items: (i) search for sensation of vice, tightness, heaviness, (ii) search for sensation of digestive or bladder spasm, (iii) pelvic floor muscle tension Individual item of DN4 pain questionnaire. Individual VAS assessing the maximum pain in the 3 months preceding the MRI, on :
  * dysmenorrhea
  * deep dyspareunia
  * non-cyclic chronic pelvic pains
  * digestive pains
  * urinary pains
VAS for pain assessement at the end of MRI-based diffusion tensor sequence, in patients with vs without endometriosis | Between 7 and 60 days after inclusion
  VAS stands for "Visual Analog Scale". The higher the worse between 0 and 10.
  MRI stands for "Magnetic Resonance Imaging".
Total examination duration and MRI-based sequence acquisition duration, in patients with vs without endometriosis | Between 7 and 60 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Louis Marcellin, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - C01 - Cochin Port Royal, Paris
  - C02-HEGP gynecology, Paris
  - C03- HEGP radiology, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision. Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).